CLINICAL TRIAL: NCT05193825
Title: Evaluation of a Visual-Analog Scale (VAS) for Remote DBS Programming
Brief Title: Evaluation of Remote DBS Programming.
Acronym: REMOTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Köglsperger (Other)
Collaborators: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other); Universitätsklinikum Leipzig (Other); Heinrich-Heine University, Duesseldorf (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital Muenster (Other)
Responsible Party: Sponsor-Investigator, Thomas Köglsperger, Resident Physician; Postdoctoral Research Fellow, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Remote DBS Programming
Record Dates: First submitted 2021-12-21; First posted 2022-01-18 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Deep Brain Stimulation; Telemedicine; Parkinson Disease
Keywords: Deep Brain Stimulation; Telemedicine; Parkinson's Disease (PD); Subthalamic Nucleus (STN); Remote
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (Active Comparator): Patients in Group A (active comparator) will have their internal pulse generator (IPG) adjusted by conventional procedures, i.e. by regular visits at their caregivers hospital.
  Interventions: Device: Standard Programming
- Group B (Experimental): Patients in Group B (experimental) will have their internal pulse generator (IPG) adjusted by using a novel software (Abbot NeurosphereTM Virtual Clinics) that allows for remote IPG programming and with the aid of a visual analogue scale (VAS).
  Interventions: Device: Remote Programming

INTERVENTIONS:
Device: Remote Programming — Patients in the experimental group (Group B) will have their internal pulse generators (IPGs) adjusted through a novel software that allows for remote DBS programming (NeurosphereTM Virtual Clinic)
  Arms: Group B
Device: Standard Programming — Patients in the active comparator group (Group A) will have their internal pulse generators (IPGs) adjusted through a standard procedure at their caregivers institution.
  Arms: Group A

SUMMARY:
Deep brain stimulation (DBS) represents the treatment of choice for advanced stages of Parkinson's disease (PD). Currently, adaptive closed-loop stimulation systems that apply disease-specific biomarkers, such as local field potentials (LFPs), are being actively examined to facilitate DBS programming. However, the most suitable feedback signal, still remains to be determined. The investigators previously tested the usefulness of the patient's subjective rating on a visual analogue scale (VAS) as a potential feedback signal for DBS adjustment and found that VAS-based programming lead to similar results as our standard approach. One of the practical advantages of using VAS-based programming strategies - in addition to saving time - is the principal applicability of such an approach to a remote programming setting, although a validation of such an approach is required. Within the scope of a prospective, randomized multicenter clinical trial (the REMOTE Trial), the investigators will examine the effectiveness and safety of VAS-based remote DBS programming in PD by using a novel and recently introduced software platform (Abbott NeurosphereTM Virtual Clinic) that allows for the programming through a smartphone-based video connection with the patient. Therefore, n = 50 PD patients undergoing STN-DBS surgery will be randomized and subsequent to surgery will have their IPG settings adjusted either during regular visits at the hospital or alternatively be programmed remotely through a VAS-based approach. Prior to surgery and after a 90 days follow-up period, we will assess specific clinical (MDS-Unified Parkinson's Disease Rating Scale = UPDRS, Parkinson's Disease Questionnaire-39 sum index = PDQ-39 SI, Beck Depression Inventory = BDI, Montreal Cognitive Assessment Scale = MOCA) parameters to determine the effectivity and safety of the two different strategies on the patient outcome and to correlate it with VAS ratings and MRI data. The results will support the examination of remote-based DBS programming and evaluate the patient's subjective judgment as a valid feedback signal.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 and 80 yrs.
* Ability to communicate with the study physician and to understand the requirements of the study
* Idiopathic Parkinson's Syndrome; IPS (according to MDS-Criteria)
* Implantation of a DBS device for the stimulation of the subthalamic nucleus (STN) to treat PD.

Exclusion Criteria:

* Any inability to communicate with the study physician and to understand the requirements of the study
* Exclusion criteria of an idiopathic Parkinson's syndrome (IPS)
* Fulfills the criteria of dementia (according to the International Classification of Diseases (ICD) 10)

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Change in UPDRS-III (Stimulation ON/Medication ON = STIM-ON/MED-ON) | Assessed at Day 90
  Part III of the MDS-Unified Parkinson's Disease Rating Scale (Range 0-128 pts. with high values indicating a more severe disease symptoms)

SECONDARY OUTCOMES:
Change in UPDRS-I | Assessed at day -1 and +90 (day 0 = implantation of DBS electrodes)
  Part I of the MDS-Parkinson's Disease Rating Scale (Range 0-52 pts. with high values indicating more severe disease symptoms)
Change in UPDRS-II | Assessed at day -1 and +90 (day 0 = implantation of DBS electrodes)
  Part II of the MDS-Parkinson's Disease Rating Scale (Range 0-52 pts. with high values indicating more severe disease symptoms)
Change in UPDRS-IV | Assessed at day -1 and +90 (day 0 = implantation of DBS electrodes)
  Part IV of the MDS-Parkinson's Disease Rating Scale (Range 0-24 pts. with high values indicating more severe disease symptoms)
Change in PDQ-39-SI | Assessed at day -1 and +90 (day 0 = implantation of DBS electrodes)
  Parkinson's Disease Questionnaire-39 Sum Index (Range 0-100 pts. with high values indicating more severe disease symptoms)
Change in Patient Rating (Patient Diary) | Assessed on a weekly basis by the patient between day +5 and +90 (day 0 = implantation of DBS electrodes)
  Number of hours spent with bothersome dyskinesia or in a reduced mobility state (OFF)
Number of visits at the the hospital or remotely | Assessed at day +90 (day 0 = implantation of DBS electrodes)
  Number of doctor-patient contacts either in person at the hospital (Group A) or remotely (Group B)
Change in TEED | Assessed at day +5 and +90 (day 0 = implantation of DBS electrodes)
  Total Electrical Energy Delivered by the IPG; TEED (1s) = (voltage2 × frequency × pulsewidth) / impedance (1s)

CONTACTS AND LOCATIONS:
Locations (1):
- Ludwig Maximilian University Hospital, Munich, Bavaria, Germany